CLINICAL TRIAL: NCT05880927
Title: Pyrotinib After Trastuzumab-based Adjuvant Therapy in Patients With HER2-positive Breast Cancer: an Open-label, Multi-center Trial
Brief Title: Pyrotinib After Trastuzumab-based Adjuvant Therapy in Patients With HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, Chief Physician, Taizhou Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERSIST
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib 400mg/day (Experimental): High risk HER2 positive patients receive pyrotinib 400mg/day for half or one year
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Patients receive pyrotinib 400mg/day for half or one year

SUMMARY:
This trial is a multicenter, open-label, phase II trial conducted at 23 centers in China. High-risk HER2 positive patients receive pyrotinib 400mg/day for one year or half year for extented adjuvant therapy.

DETAILED DESCRIPTION:
Patients must meet one of the following criteria: N stage ≥1; T stage ≥2; did not achieve pathological complete response (pCR) after neoadjuvant therapy; had pCR after neoadjuvant therapy but with tumor size ≥ 5cm or N stage ≥2; or tumor size less than 2cm but with high Ki67; histologic grade 3 or with lymph node micrometastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-75 years old
2. HER2 positive breast cancer
3. ECOG PS 0-1
4. Known hormone receptor status
5. Completed 1 year of trastuzumab-based adjuvant therapy within 6 months
6. Patients at high risk

Exclusion Criteria:

1. Serious heart disease or discomfort
2. Inability to swallow, intestinal obstruction, or the presence of other factors that interfere with drug administration and absorption
3. Known allergic history of drug components of this regimen
4. A history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation
5. Pregnant and lactating female patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
iDFS | From date of receiving drug until the date of first documented invasive disease or date of death from any cause, whichever came first, assessed up to 60 months
  INVASIVE DISEASE FREE SURVIVAL

SECONDARY OUTCOMES:
OS | From date of receiving drug until the date of death from any cause, assessed up to 60 months
  Overall Survival
Adverse events | through study completion, an average of 5 years
  frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Feilin Cao, Master, Principal Investigator — Taizhou Hospital
Locations (1):
- Taizhou Hospital, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao F, Ma Z, Wu Z, Wu W, Wang O, Cui B, Zhu X, Hao J, Ji X, Li Z, Tao D, Feng Q, Lin W, Shi D, Shu J, Zhou J, Huang S. Pyrotinib after trastuzumab-based adjuvant therapy in patients with HER2-positive breast cancer (PERSIST): A multicenter phase II trial. Elife. 2025 Apr 3;13:RP101724. doi: 10.7554/eLife.101724. PMID 40178527